CLINICAL TRIAL: NCT00372593
Title: A Phase III Randomized Trial of Gemtuzumab Ozogamicin (Mylotarg) Combined With Conventional Chemotherapy for De Novo Acute Myeloid Leukemia (AML) in Children, Adolescents, and Young Adults
Brief Title: Combination Chemotherapy With or Without Gemtuzumab in Treating Young Patients With Newly Diagnosed Acute Myeloid Leukemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAML0531; COG-AAML0531 (Other: Children's Oncology Group); CDR0000487497 (Other: Clinical Trials.gov); NCI-2009-00320 (Registry Identifier: Clinical Trials Reporting Program)
Record Dates: First submitted 2006-09-06; First posted 2006-09-07 (Estimated); Results first posted 2015-01-13 (Estimated); Last update posted 2021-03-24 (Actual); Status verified 2017-02

CONDITIONS: Leukemia
Keywords: adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); untreated adult acute myeloid leukemia; untreated childhood acute myeloid leukemia and other myeloid malignancies; adult acute basophilic leukemia; adult acute eosinophilic leukemia; adult acute minimally differentiated myeloid leukemia (M0); adult acute myeloblastic leukemia without maturation (M1); adult acute myeloblastic leukemia with maturation (M2); adult acute myelomonocytic leukemia (M4); adult acute monoblastic leukemia (M5a); adult acute monocytic leukemia (M5b); adult erythroleukemia (M6a); adult pure erythroid leukemia (M6b); adult acute megakaryoblastic leukemia (M7); childhood acute basophilic leukemia; childhood acute eosinophilic leukemia; childhood acute minimally differentiated myeloid leukemia (M0); childhood acute myeloblastic leukemia without maturation (M1); childhood acute myeloblastic leukemia with maturation (M2); childhood acute myelomonocytic leukemia (M4); childhood acute monocytic leukemia (M5b); childhood acute monoblastic leukemia (M5a); childhood acute erythroleukemia (M6); childhood acute megakaryocytic leukemia (M7)
MeSH Terms: conditions — Leukemia; Congenital Abnormalities; Leukemia, Basophilic, Acute; Leukemia, Eosinophilic, Acute; Leukemia, Myeloid, Acute; Leukemia, Myelomonocytic, Acute; Leukemia, Monocytic, Acute; Leukemia, Erythroblastic, Acute; Leukemia, Megakaryoblastic, Acute | interventions — Asparaginase; Cytarabine; Daunorubicin; Etoposide; etoposide phosphate; Gemtuzumab; Mitoxantrone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm A: Standard Arm - No GMTZ, AML Pts w/out Down Syndrome (Active Comparator): Patients receive intrathecal (IT) cytarabine (ARA-C) at diagnosis or on day 1 of treatment or twice a week for up to 6 doses. They also receive an infusion of ARA-C on days 1-10; a 6-hour infusion of daunorubicin hydrochloride on days 1, 3, and 5; and a 4-hr infusion of etoposide on days 1-5.
  After 3 weeks of rest, patients receive IT ARA-C on day 1. They also receive an infusion of ARA-C on days 1-8; a 6-hr infusion of daunorubicin on days 1, 3, and 5; and a 4-hr infusion of etoposide on days 1-5.
  After 3 weeks of rest, some patients receive IT ARA-C on day 1 and 1-hr infusions of ARA-C and etoposide on days 1-5.
  After 3 weeks of rest, some patients receive IT ARA-C on day 1; a 2-hr infusion of ARA-C on days 1-4; and a 1-hour infusion of mitoxantrone on days 3-6. After 3 weeks of rest, they receive a 3-hr infusion of ARA-C on days 1, 2, 8, and 9 and an injection of asparaginase on days 2 and 9.
  Interventions: Drug: asparaginase; Drug: cytarabine; Drug: daunorubicin hydrochloride; Drug: etoposide; Drug: mitoxantrone hydrochloride
- Arm B: Experimental - with GMTZ, AML Pts w/out Down Syndrome (Experimental): Pts receive IT ARA-C at diagnosis or on day 1 of treatment or twice a week for up to six doses. They also receive an infusion of ARA-C on days 1-10; a 6-hr infusion of daunorubicin on days 1, 3, & 5; a 4-hr infusion of etoposide on days 1-5; and a 2-hr infusion of GMTZ - gemtuzumab ozogamicin (Mylotarg) on day 6. After 3 wks of rest, patients receive IT ARA-C on day 1. They also receive an infusion of ARA-C on days 1-8; a 6-hr infusion of daunorubicin on days 1, 3, and 5; and a 4-hr infusion of etoposide on days 1-5. After 3 weeks of rest, some patients receive IT ARA-C on day 1 and 1-hr infusions of ARA-C and etoposide on days 1-5. After 3 wks of rest, some patients receive IT ARA-C on day 1; a 2-hr infusion of ARA-C on days 1-4; and a 1-hr infusion of mitoxantrone hydrochloride on days 3-6. They also receive a 2-hr infusion of gemtuzumab on day 7. After 3 weeks of rest, they receive a 3-hr infusion of ARA-C on days 1, 2, 8, and 9 and an injection of asparaginase on days 2 and 9.
  Interventions: Drug: asparaginase; Drug: cytarabine; Drug: daunorubicin hydrochloride; Drug: etoposide; Drug: gemtuzumab ozogamicin; Drug: mitoxantrone hydrochloride
- Arm A: Standard Arm - No GMTZ, AML Patients with Down Syndrome (Active Comparator): Patients receive intrathecal (IT) cytarabine (ARA-C) at diagnosis or on day 1 of treatment or twice a week for up to 6 doses. They also receive an infusion of ARA-C on days 1-10; a 6-hour infusion of daunorubicin hydrochloride on days 1, 3, and 5; and a 4-hr infusion of etoposide on days 1-5.
  After 3 weeks of rest, patients receive IT ARA-C on day 1. They also receive an infusion of ARA-C on days 1-8; a 6-hr infusion of daunorubicin on days 1, 3, and 5; and a 4-hr infusion of etoposide on days 1-5.
  After 3 weeks of rest, some patients receive IT ARA-C on day 1 and 1-hr infusions of ARA-C and etoposide on days 1-5.
  After 3 weeks of rest, some patients receive IT ARA-C on day 1; a 2-hr infusion of ARA-C on days 1-4; and a 1-hour infusion of mitoxantrone on days 3-6. After 3 weeks of rest, they receive a 3-hr infusion of ARA-C on days 1, 2, 8, and 9 and an injection of asparaginase on days 2 and 9.
  Interventions: Drug: asparaginase; Drug: cytarabine; Drug: daunorubicin hydrochloride; Drug: etoposide; Drug: mitoxantrone hydrochloride

INTERVENTIONS:
Drug: asparaginase — Given intramuscularly
  Other Names: E.coli; E.coli L-asparaginase; EC 3.5.2.2; colaspase; L-asnase; Elspar; Kidrolase; Crasnitin; Leunase; NSC 109229
Drug: cytarabine — Given IV
  Other Names: Cytosine arabinoside; Ara-C; Cytosar; NSC # 63878
Drug: daunorubicin hydrochloride — Given IV over 6 hours
  Other Names: Daunomycin; rubidomycin; Cerubidine; NSC #82151
Drug: etoposide — Given IV over 1-4 hours
  Other Names: VePesid; Etopophos; VP-16; NSC #141540
Drug: gemtuzumab ozogamicin — Given IV over 2 hours
  Other Names: Mylotarg; GMTZ
  Arms: Arm B: Experimental - with GMTZ, AML Pts w/out Down Syndrome
Drug: mitoxantrone hydrochloride — Given IV over 1 hour
  Other Names: Novantrone; CL 232315; DAD; DHAD; Mitozantrone; NSC #301739

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as gemtuzumab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Giving combination chemotherapy together with gemtuzumab may kill more cancer cells. It is not yet known whether combination chemotherapy is more effective with or without gemtuzumab in treating patients with newly diagnosed acute myeloid leukemia.

PURPOSE: This randomized phase III trial is studying combination chemotherapy and gemtuzumab to see how well they work compared with combination chemotherapy alone in treating young patients with newly diagnosed acute myeloid leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the event-free survival (EFS) and overall survival (OS) of young patients with newly diagnosed acute myeloid leukemia (AML) treated with conventional combination chemotherapy with vs without gemtuzumab ozogamicin (GMTZ).

Secondary

* Compare the remission induction rates after two courses of therapy in these patients.
* Compare disease-free survival and OS in patients who are eligible for an human leukocyte antigen (HLA)-matched family donor (MFD) stem cell transplant (SCT) by virtue of their risk classification, with patients assigned to MFD SCT if a MFD is available, or to chemotherapy if a MFD is not available.
* Determine the outcome of patients with Down syndrome who are 4 years of age or older at diagnosis and treated with conventional combination chemotherapy without GMTZ.
* Compare the EFS and OS of patients with de novo AML treated with conventional combination chemotherapy with vs without GMTZ censoring MFD SCT recipients.
* Determine the prevalence and prognostic significance of molecular abnormalities of KIT, CCAAT-enhancer binding protein alpha (CEBPα) and MLL-Partial tandem duplications (PTD) genes in these patients.
* Determine the leukemic involvement of hematopoietic early progenitor and its role in defining response to therapy.
* Assess the ability of a second-generation flow cytometric assay to predict patients at high risk for relapse during periods of clinical remission.
* Examine whether GMTZ significantly improves EFS and OS in patients with higher CD33 concentrations/intensity.
* Examine whether GMTZ significantly improves complete remission, EFS, and OS in each of the cytogenetic risk groups (high-, intermediate-, and low-risk) identified in prior Medical Research Council trials.
* Utilize fluorescence in situ hybridization (FISH) analysis to identify variant patterns among subgroups of patients who demonstrate the same G-banded chromosomal abnormality (e.g., inv[16]/t[16;16], t[8;21], 11q23 abnormality) and determine whether these variant patterns account for the heterogeneity of responses to therapy.
* Examine the impact of complex karyotypes (≥ 3, ≥ 4, and ≥ 5 abnormalities) on OS and EFS in intermediate-risk patients for whom no high-risk or low-risk cytogenetic abnormalities exist.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to relapse risk (high vs intermediate vs low). Patients are randomized to 1 of 2 treatment arms. Patients with Down syndrome are nonrandomly assigned to arm I (but do not undergo allogeneic stem cell transplant [SCT]).

* Arm I (standard therapy):

  * Induction 1: Patients receive cytarabine IT at the time of diagnosis or on day 1*. Patients also receive cytarabine IV on days 1-10, daunorubicin hydrochloride IV over 6 hours on days 1, 3, and 5, and etoposide IV over 4 hours on days 1-5. After 3 weeks of rest, all patients (regardless of remission status) proceed to induction 2.

NOTE: *Patients with Central Nervous System (CNS) disease receive cytarabine IT twice weekly until the cerebrospinal fluid is clear, followed by two additional IT treatments. Patients with refractory CNS leukemia after 6 doses of IT treatment are removed from the study.

* Induction 2: Patients receive cytarabine IT on day 1, cytarabine IV on days 1-8, daunorubicin hydrochloride IV over 6 hours on days 1, 3, and 5, and etoposide IV over 4 hours on days 1-5. After 3 weeks of rest, patients in complete remission (CR) proceed to intensification 1. Patients with refractory disease are removed from protocol therapy.
* Intensification 1: Patients receive cytarabine IT on day 1, high-dose cytarabine IV over 1 hour on days 1-5, and etoposide IV over 1 hour on days 1-5. After 3 weeks of rest, patients in remission proceed to intensification 2, followed by intensification 3. Patients in remission proceed to allogeneic SCT 2-8 weeks after blood counts recover. Patients with high-risk disease with an alternative donor proceed to intensification 2 and 3, followed by allogeneic SCT. Patients not in remission are removed from protocol therapy.
* Intensification 2: Patients receive cytarabine IT on day 1, high-dose cytarabine IV over 2 hours on days 1-4, and mitoxantrone hydrochloride IV over 1 hour on days 3-6. After 3 weeks of rest, patients proceed to intensification 3.
* Intensification 3: Patients receive high-dose cytarabine IV over 3 hours on days 1, 2, 8, and 9 and asparaginase intramuscularly on days 2 and 9.

  * Arm II:
* Induction 1: Patients receive treatment as in induction 1 of arm I. Patients also receive gemtuzumab ozogamicin (GMTZ) IV over 2 hours on day 6.
* Induction 2: Patients receive treatment as in induction 2 of arm I.
* Intensification 1: Patients receive treatment as in intensification 1 of arm I.
* Intensification 2: Patients receive treatment as in intensification 2 of arm I. Patients also receive GMTZ IV over 2 hours on day 7.
* Intensification 3: Patients receive treatment as in intensification 3 of arm I.

  * Allogeneic SCT (for patients with intermediate- or high-risk disease):
* MFD: Patients receive a conditioning regimen comprising busulfan IV over 2 hours every 6 hours on days -9 to -6 and cyclophosphamide IV over 1 hour on days -5 to -2. Patients undergo allogeneic SCT on day 0. Patients receive cyclosporine IV or orally twice daily on days -1 to 180 and methotrexate IV on days 1, 3, 6, and 11. Patients receive graft-vs-host disease (GVHD) prophylaxis comprising cyclosporine IV over 1-4 hours or orally twice daily on days -1 to 180 and methotrexate IV on days 1, 3, 6, and 11.
* Matched alternative donor: Patients receive a conditioning regimen comprising busulfan and cyclophosphamide as above. Patients also receive antithymocyte globulin IV over 6-8 hours on days -3 to -1. Patients then undergo allogeneic SCT and receive GVHD prophylaxis as above.

After completion of study treatment, patients are followed periodically for 3 years and then annually thereafter.

PROJECTED ACCRUAL: A total of 1,012 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Newly diagnosed acute myeloid leukemia (AML)

  * Meets customary criteria for AML with ≥ 20% bone marrow blasts (by WHO classification)

    * Patients with < 20% bone marrow blasts and cytopenia or myelodysplastic syndromes (e.g., chronic myelomonocytic leukemia, refractory anemia (RA), RA with excess blasts, RA with ringed sideroblasts) are eligible provided 1 of the following criteria is met:

      * Karyotypic abnormality characteristic of de novo AML (t[8;21][q22;q22], inv[16][p13q22], t[16;16][p13;q22], or 11q23 abnormalities)
      * Unequivocal presence of megakaryoblasts (by WHO classification)
  * Isolated myeloid sarcoma (i.e., myeloblastoma or chloroma) allowed regardless of bone marrow results
* Infants < 1 month of age with progressive disease* are eligible NOTE: *Infants < 1 month of age with AML may be given supportive care until it is clear that the leukemia is not regressing (i.e., the disappearance of peripheral blasts and the normalization of peripheral blood counts)
* Patients with Down syndrome ≥ 4 years of age are eligible
* No juvenile myelomonocytic leukemia
* No Fanconi's anemia, Kostmann syndrome, Shwachman syndrome, or any other known bone marrow failure syndrome
* No promyelocytic leukemia (M3)
* No secondary or treatment-related AML
* Matched family donor criteria (for patients with intermediate-risk or high-risk disease):

  * HLA-A, -B, -C, and beta chain (-DRB1), identical or 1 antigen or allele mismatched by molecular high resolution technique
  * All available first-degree family members (parents and siblings) must be HLA typed
  * No syngeneic donors
* Matched alternative donor criteria (for patients with high-risk disease):

  * HLA-A, -B, -C, and -DRB1, identical or 1 antigen or allele mismatched donor
  * HLA-A, -B, and -DRB1 4 of 6 antigen matched unrelated cord blood donor
  * Mismatched family member donor with ≥ 1 haplotype match or 5 of 6 antigen phenotypic match

PATIENT CHARACTERISTICS:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy, radiation therapy, or any antileukemic therapy

  * Topical or inhalation steroids for other conditions allowed
  * Intrathecal cytarabine given at diagnosis allowed
* No other prior treatment for AML
* No concurrent peripheral blood stem cell transplantation in patients with matched family donor

Max Age: 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1070 (Actual)
Dates: Start 2006-08; Primary Completion 2013-08 (Actual); Study Completion 2020-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan S. Gamis, MD, MPH, Study Chair — Children's Mercy Hospital Kansas City; Richard Aplenc, MD, MSCE, Study Chair — Children's Hospital of Philadelphia
Locations (198):
- United States (178):
  - UAB Comprehensive Cancer Center, Birmingham, Alabama
  - University of South Alabama Mitchell Cancer Institute, Mobile, Alabama
  - Banner Desert Medical Center, Mesa, Arizona
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Arizona Cancer Center at University of Arizona Health Sciences Center, Tucson, Arizona
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Southern California Permanente Medical Group, Downey, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Loma Linda University Cancer Institute at Loma Linda University Medical Center, Loma Linda, California
  - Childrens Hospital Los Angeles, Los Angeles, California
  - Samuel Oschin Comprehensive Cancer Institute at Cedars-Sinai Medical Center, Los Angeles, California
  - Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California
  - Children's Hospital Central California, Madera, California
  - Children's Hospital and Research Center Oakland, Oakland, California
  - Kaiser Permanente Medical Center - Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Sutter Cancer Center, Sacramento, California
  - University of California Davis Cancer Center, Sacramento, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Santa Barbara Cottage Children's Hospital, Santa Barbara, California
  - Jonathan Jaques Children's Cancer Center at Miller Children's Hospital, Torrance, California
  - Children's Hospital Center for Cancer and Blood Disorders, Aurora, Colorado
  - Carole and Ray Neag Comprehensive Cancer Center at the University of Connecticut Health Center, Farmington, Connecticut
  - Yale Cancer Center, New Haven, Connecticut
  - Alfred I. duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Broward General Medical Center Cancer Center, Fort Lauderdale, Florida
  - Lee Cancer Care of Lee Memorial Health System, Fort Myers, Florida
  - University of Florida Shands Cancer Center, Gainesville, Florida
  - Memorial Cancer Institute at Memorial Regional Hospital, Hollywood, Florida
  - Nemours Children's Clinic, Jacksonville, Florida
  - University of Miami Sylvester Comprehensive Cancer Center - Miami, Miami, Florida
  - Miami Children's Hospital, Miami, Florida
  - Baptist-South Miami Regional Cancer Program, Miami, Florida
  - Florida Hospital Cancer Institute at Florida Hospital Orlando, Orlando, Florida
  - M.D. Anderson Cancer Center at Orlando, Orlando, Florida
  - Nemours Children's Clinic - Orlando, Orlando, Florida
  - Sacred Heart Cancer Center at Sacred Heart Hospital, Pensacola, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - St. Joseph's Cancer Institute at St. Joseph's Hospital, Tampa, Florida
  - Kaplan Cancer Center at St. Mary's Medical Center, West Palm Beach, Florida
  - AFLAC Cancer Center and Blood Disorders Service of Children's Healthcare of Atlanta - Egleston Campus, Atlanta, Georgia
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - MBCCOP - Medical College of Georgia Cancer Center, Augusta, Georgia
  - Curtis and Elizabeth Anderson Cancer Institute at Memorial Health University Medical Center, Savannah, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - Tripler Army Medical Center, Tripler AMC, Hawaii
  - Mountain States Tumor Institute at St. Luke's Regional Medical Center, Boise, Idaho
  - University of Illinois Cancer Center, Chicago, Illinois
  - Children's Memorial Hospital - Chicago, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Keyser Family Cancer Center at Advocate Hope Children's Hospital, Oak Lawn, Illinois
  - Advocate Lutheran General Cancer Care Center, Park Ridge, Illinois
  - Simmons Cooper Cancer Institute, Springfield, Illinois
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - St. Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Kansas Masonic Cancer Research Institute at the University of Kansas Medical Center, Kansas City, Kansas
  - Lucille P. Markey Cancer Center at University of Kentucky, Lexington, Kentucky
  - Kosair Children's Hospital, Louisville, Kentucky
  - Tulane Cancer Center Office of Clinical Research, Alexandria, Louisiana
  - Children's Hospital of New Orleans, New Orleans, Louisiana
  - CancerCare of Maine at Eastern Maine Medical Center, Bangor, Maine
  - Maine Children's Cancer Program at Barbara Bush Children's Hospital, Portland, Maine
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - Alvin and Lois Lapidus Cancer Institute at Sinai Hospital, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Floating Hospital for Children at Tufts - New England Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - Baystate Regional Cancer Program at D'Amour Center for Cancer Care, Springfield, Massachusetts
  - UMASS Memorial Cancer Center - University Campus, Worcester, Massachusetts
  - C.S. Mott Children's Hospital at University of Michigan Medical Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Butterworth Hospital at Spectrum Health, Grand Rapids, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - Breslin Cancer Center at Ingham Regional Medical Center, Lansing, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - Masonic Cancer Center at University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - University of Mississippi Cancer Clinic, Jackson, Mississippi
  - Ellis Fischel Cancer Center at University of Missouri - Columbia, Columbia, Missouri
  - Children's Mercy Hospital, Kansas City, Missouri
  - Cardinal Glennon Children's Hospital, St Louis, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - Children's Hospital, Omaha, Nebraska
  - UNMC Eppley Cancer Center at the University of Nebraska Medical Center, Omaha, Nebraska
  - CCOP - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Hackensack University Medical Center Cancer Center, Hackensack, New Jersey
  - Cancer Institute of New Jersey at UMDNJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - St. Joseph's Hospital and Medical Center, Paterson, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Albany Medical Center Hospital, Albany, New York
  - Brooklyn Hospital Center, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Winthrop University Hospital, Mineola, New York
  - Schneider Children's Hospital, New Hyde Park, New York
  - NYU Cancer Institute at New York University Medical Center, New York, New York
  - New York Weill Cornell Cancer Center at Cornell University, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - Herbert Irving Comprehensive Cancer Center at Columbia University Medical Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Stony Brook University Cancer Center, Stony Brook, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Albert Einstein Cancer Center at Albert Einstein College of Medicine, The Bronx, New York
  - Mission Hospitals - Memorial Campus, Asheville, North Carolina
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Presbyterian Cancer Center at Presbyterian Hospital, Charlotte, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Leo W. Jenkins Cancer Center at ECU Medical School, Greenville, North Carolina
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - Akron Children's Hospital, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Medical Center - Dayton, Dayton, Ohio
  - Toledo Hospital, Toledo, Ohio
  - Medical University of Ohio Cancer Center, Toledo, Ohio
  - Oklahoma University Cancer Institute, Oklahoma City, Oklahoma
  - Legacy Emanuel Hospital and Health Center and Children's Hospital, Portland, Oregon
  - Knight Cancer Institute at Oregon Health and Science University, Portland, Oregon
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Geisinger Cancer Institute at Geisinger Health, Danville, Pennsylvania
  - Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St. Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Rhode Island Hospital Comprehensive Cancer Center, Providence, Rhode Island
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - Palmetto Health South Carolina Cancer Center, Columbia, South Carolina
  - Greenville Hospital Cancer Center, Greenville, South Carolina
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - T.C. Thompson Children's Hospital, Chattanooga, Tennessee
  - East Tennessee Children's Hospital, Knoxville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Texas Tech University Health Sciences Center School of Medicine - Amarillo, Amarillo, Texas
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - Simmons Comprehensive Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - Cook Children's Medical Center - Fort Worth, Fort Worth, Texas
  - Baylor University Medical Center - Houston, Houston, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Primary Children's Medical Center, Salt Lake City, Utah
  - Fletcher Allen Health Care - University Health Center Campus, Burlington, Vermont
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Naval Medical Center - Portsmouth, Portsmouth, Virginia
  - Virginia Commonwealth University Massey Cancer Center, Richmond, Virginia
  - Carilion Medical Center for Children at Roanoke Community Hospital, Roanoke, Virginia
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington
  - Providence Cancer Center at Sacred Heart Medical Center, Spokane, Washington
  - Mary Bridge Children's Hospital and Health Center - Tacoma, Tacoma, Washington
  - Madigan Army Medical Center - Tacoma, Tacoma, Washington
  - West Virginia University Health Sciences Center - Charleston, Charleston, West Virginia
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - University of Wisconsin Paul P. Carbone Comprehensive Cancer Center, Madison, Wisconsin
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin
  - Midwest Children's Cancer Center at Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Australia (4):
  - Westmead Institute for Cancer Research at Westmead Hospital, Westmead, New South Wales
  - Royal Children's Hospital, Herston, Queensland
  - Women's and Children's Hospital, North Adelaide, South Australia
  - Princess Margaret Hospital for Children, Perth, Western Australia
- Canada (11):
  - Children's & Women's Hospital of British Columbia, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Janeway Children's Health and Rehabilitation Centre, St. John's, Newfoundland and Labrador
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Cancer Centre of Southeastern Ontario at Kingston General Hospital, Kingston, Ontario
  - Children's Hospital of Western Ontario, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - Hopital Sainte Justine, Montreal, Quebec
  - Centre Hospitalier Universitaire de Quebec, Québec
- New Zealand (2):
  - Christchurch Hospital, Christchurch
  - Starship Children's Health, Grafton
- San Jorge Children's Hospital, Santurce, Puerto Rico
- Switzerland (2):
  - Swiss Pediatric Oncology Group Bern, Bern
  - Swiss Pediatric Oncology Group Geneva, Geneva

REFERENCES:
- [Background] Pollard JA, Alonzo TA, Loken M, Gerbing RB, Ho PA, Bernstein ID, Raimondi SC, Hirsch B, Franklin J, Walter RB, Gamis A, Meshinchi S. Correlation of CD33 expression level with disease characteristics and response to gemtuzumab ozogamicin containing chemotherapy in childhood AML. Blood. 2012 Apr 19;119(16):3705-11. doi: 10.1182/blood-2011-12-398370. Epub 2012 Feb 29. PMID 22378848
- [Result] Gamis AS, Alonzo TA, Meshinchi S, Sung L, Gerbing RB, Raimondi SC, Hirsch BA, Kahwash SB, Heerema-McKenney A, Winter L, Glick K, Davies SM, Byron P, Smith FO, Aplenc R. Gemtuzumab ozogamicin in children and adolescents with de novo acute myeloid leukemia improves event-free survival by reducing relapse risk: results from the randomized phase III Children's Oncology Group trial AAML0531. J Clin Oncol. 2014 Sep 20;32(27):3021-32. doi: 10.1200/JCO.2014.55.3628. PMID 25092781
- [Derived] Huang BJ, Meyer LK, Alonzo TA, Wang YC, Lamble AJ, Ries RE, Wang W, Hirsch B, Raca G, Ma X, Gamis AS, Aplenc R, Kolb EA, Cooper TM, Tarlock K, Loken MR, Meshinchi S, Chewning JH, Woods WG, Horan JT. Hematopoietic Stem Cell Transplantation Outcomes for High-Risk AML: A Report From the Children's Oncology Group. J Clin Oncol. 2025 Jun 10;43(17):1961-1971. doi: 10.1200/JCO-24-01841. Epub 2025 Apr 28. PMID 40294366
- [Derived] Tarlock K, Gerbing RB, Ries RE, Smith JL, Leonti A, Huang BJ, Kirkey D, Robinson L, Peplinski JH, Lange B, Cooper TM, Gamis AS, Kolb EA, Aplenc R, Pollard JA, Alonzo TA, Meshinchi S. Prognostic impact of cooccurring mutations in FLT3-ITD pediatric acute myeloid leukemia. Blood Adv. 2024 May 14;8(9):2094-2103. doi: 10.1182/bloodadvances.2023011980. PMID 38295280
- [Derived] Zarnegar-Lumley S, Alonzo TA, Gerbing RB, Othus M, Sun Z, Ries RE, Wang J, Leonti A, Kutny MA, Ostronoff F, Radich JP, Appelbaum FR, Pogosova-Agadjanyan EL, O'Dwyer K, Tallman MS, Litzow M, Atallah E, Cooper TM, Aplenc RA, Abdel-Wahab O, Gamis AS, Luger S, Erba H, Levine R, Kolb EA, Stirewalt DL, Meshinchi S, Tarlock K. Characteristics and prognostic impact of IDH mutations in AML: a COG, SWOG, and ECOG analysis. Blood Adv. 2023 Oct 10;7(19):5941-5953. doi: 10.1182/bloodadvances.2022008282. PMID 37267439
- [Derived] Bertrums EJM, Smith JL, Harmon L, Ries RE, Wang YJ, Alonzo TA, Menssen AJ, Chisholm KM, Leonti AR, Tarlock K, Ostronoff F, Pogosova-Agadjanyan EL, Kaspers GJL, Hasle H, Dworzak M, Walter C, Muhlegger N, Morerio C, Pardo L, Hirsch B, Raimondi S, Cooper TM, Aplenc R, Gamis AS, Kolb EA, Farrar JE, Stirewalt D, Ma X, Shaw TI, Furlan SN, Brodersen LE, Loken MR, Van den Heuvel-Eibrink MM, Zwaan CM, Triche TJ, Goemans BF, Meshinchi S. Comprehensive molecular and clinical characterization of NUP98 fusions in pediatric acute myeloid leukemia. Haematologica. 2023 Aug 1;108(8):2044-2058. doi: 10.3324/haematol.2022.281653. PMID 36815378
- [Derived] Elgarten CW, Wood AC, Li Y, Alonzo TA, Brodersen LE, Gerbing RB, Getz KD, Huang YV, Loken M, Meshinchi S, Pollard JA, Sung L, Woods WG, Kolb EA, Gamis AS, Aplenc R. Outcomes of intensification of induction chemotherapy for children with high-risk acute myeloid leukemia: A report from the Children's Oncology Group. Pediatr Blood Cancer. 2021 Dec;68(12):e29281. doi: 10.1002/pbc.29281. Epub 2021 Oct 1. PMID 34596937
- [Derived] Brodersen LE, Gerbing RB, Pardo ML, Alonzo TA, Paine D, Fritschle W, Hsu FC, Pollard JA, Aplenc R, Kahwash SB, Hirsch B, Ramondi S, Wells D, Kolb EA, Gamis AS, Meshinchi S, Loken MR. Morphologic remission status is limited compared to DeltaN flow cytometry: a Children's Oncology Group AAML0531 report. Blood Adv. 2020 Oct 27;4(20):5050-5061. doi: 10.1182/bloodadvances.2020002070. PMID 33080007
- [Derived] Voigt AP, Brodersen LE, Alonzo TA, Gerbing RB, Menssen AJ, Wilson ER, Kahwash S, Raimondi SC, Hirsch BA, Gamis AS, Meshinchi S, Wells DA, Loken MR. Phenotype in combination with genotype improves outcome prediction in acute myeloid leukemia: a report from Children's Oncology Group protocol AAML0531. Haematologica. 2017 Dec;102(12):2058-2068. doi: 10.3324/haematol.2017.169029. Epub 2017 Sep 7. PMID 28883080
- [Derived] Eidenschink Brodersen L, Alonzo TA, Menssen AJ, Gerbing RB, Pardo L, Voigt AP, Kahwash SB, Hirsch B, Raimondi S, Gamis AS, Meshinchi S, Loken MR. A recurrent immunophenotype at diagnosis independently identifies high-risk pediatric acute myeloid leukemia: a report from Children's Oncology Group. Leukemia. 2016 Oct;30(10):2077-2080. doi: 10.1038/leu.2016.119. Epub 2016 May 2. No abstract available. PMID 27133823
- [Derived] Sung L, Aplenc R, Alonzo TA, Gerbing RB, Lehrnbecher T, Gamis AS. Effectiveness of supportive care measures to reduce infections in pediatric AML: a report from the Children's Oncology Group. Blood. 2013 May 2;121(18):3573-7. doi: 10.1182/blood-2013-01-476614. Epub 2013 Mar 7. PMID 23471307
- See also: Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive — https://nctn-data-archive.nci.nih.gov/

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm B: Experimental - With GMTZ, AML Pts w/Out Down Syndrome: Pts receive IT ARA-C at diagnosis or on day 1 of treatment or twice a week for up to six doses. They also receive an infusion of ARA-C on days 1-10; a 6-hr infusion of daunorubicin on days 1, 3, & 5; a 4-hr infusion of etoposide on days 1-5; and a 2-hr infusion of gemtuzumab ozogamicin (GMTZ) (Mylotarg) on day 6. After 3 wks of rest, patients receive IT ARA-C on day 1. They also receive an infusion of ARA-C on days 1-8; a 6-hr infusion of daunorubicin on days 1, 3, and 5; and a 4-hr infusion of etoposide on days 1-5. After 3 weeks of rest, some patients receive IT ARA-C on day 1 and 1-hr infusions of ARA-C and etoposide on days 1-5. After 3 wks of rest, some patients receive IT ARA-C on day 1; a 2-hr infusion of ARA-C on days 1-4; and a 1-hr infusion of mitoxantrone hydrochloride on days 3-6. They also receive a 2-hr infusion of gemtuzumab on day 7. After 3 weeks of rest, they receive a 3-hr infusion of ARA-C on days 1, 2, 8, and 9 and an injection of asparaginase on days 2 and 9.
Period: Overall Study
Arm/Group | Arm A: Standard Arm - No GMTZ, AML Pts w/Out Down Syndrome | Arm B: Experimental - With GMTZ, AML Pts w/Out Down Syndrome | Arm A: Standard Arm - No GMTZ, AML Patients With Down Syndrome
Started | 531 | 532 | 7
Completed | 327 | 334 | 3
Not Completed | 204 | 198 | 4
Not completed — Adverse Event | 43 | 45 | 0
Not completed — Death | 16 | 20 | 1
Not completed — Lack of Efficacy | 82 | 71 | 2
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Physician Decision | 42 | 41 | 0
Not completed — Ineligible | 20 | 21 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Standard Arm - No GMTZ, AML Pts w/Out Down Syndrome | Arm B: Experimental - With GMTZ, AML Pts w/Out Down Syndrome | Arm A: Standard Arm - No GMTZ, AML Patients With Down Syndrome | Total
Number analyzed (Participants) | 531 | 532 | 7 | 1070
Age, Continuous [Mean (Standard Deviation); unit: days] | 3352.86 (2336.55) | 3466 (2283.45) | 4206.71 (1979.95) | 3409.43 (2310)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 516 | 510 | 7 | 1033
  Between 18 and 65 years | 15 | 22 | 0 | 37
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 260 | 277 | 4 | 541
  Male | 271 | 255 | 3 | 529
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 1 | 0 | 4
  Asian | 28 | 24 | 0 | 52
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 0 | 2
  Black or African American | 62 | 58 | 2 | 122
  White | 383 | 394 | 5 | 782
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 54 | 54 | 0 | 108
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 100 | 97 | 0 | 197
  Not Hispanic or Latino | 411 | 416 | 7 | 834
  Unknown or Not Reported | 20 | 19 | 0 | 39
Region of Enrollment [Number; unit: participants]
  United States | 473 | 480 | 5 | 958
  Canada | 34 | 32 | 2 | 68
  Australia | 19 | 15 | 0 | 34
  Switzerland | 1 | 0 | 0 | 1
  New Zealand | 4 | 5 | 0 | 9

OUTCOME MEASURES:

1. Primary Outcome: Event-free Survival at 3 Years
Description: The Kaplan-Meier method will be used to calculate estimates of Event Free Survival (EFS). The log-rank test will be used to compare survival between treatment groups. Analysis of EFS of Down syndrome patients will be performed separately. Monitoring for efficacy of GMTZ with respect to Overall Survival (OS) and EFS will utilize monitoring based on the Lan-DeMets criterion with α-spending function αt^2 (truncated at 3 standard deviations) and 2.5% type I error.
Time Frame: Time from study entry to time of induction failure, relapse, or death, assessed at 3 years
Population: Ineligible patients are excluded from analyses of Overall Survival and Event Free Survival.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A: Standard Arm - No GMTZ, AML Pts w/Out Down Syndrome | Arm B: Experimental - With GMTZ, AML Pts w/Out Down Syndrome | Arm A: Standard Arm - No GMTZ, AML Patients With Down Syndrome
Number analyzed (Participants) | 511 | 511 | 6
percentage of participants | 46.9 [42.5 to 51.3] | 53.1 [48.6 to 57.4] | 50.0 [11.1 to 80.4]

2. Primary Outcome: Overall Survival at 3 Years
Description: The Kaplan-Meier method will be used to calculate estimates of OS. Analysis of OS of Down syndrome patients will be performed separately. Monitoring for efficacy of GMTZ with respect to OS and EFS will utilize monitoring based on the Lan-DeMets criterion with α-spending function αt^2 (truncated at 3 standard deviations) and 2.5% type I error.
Time Frame: Time from study entry, assessed at 3 years
Population: Ineligible patients are excluded from analyses of Overall Survival and Event Free Survival.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A: Standard Arm - No GMTZ, AML Pts w/Out Down Syndrome | Arm B: Experimental - With GMTZ, AML Pts w/Out Down Syndrome | Arm A: Standard Arm - No GMTZ, AML Patients With Down Syndrome
Number analyzed (Participants) | 511 | 511 | 6
percentage of participants | 65.4 [61.0 to 69.4] | 69.4 [65.1 to 73.3] | 50.0 [11.1 to 80.4]

3. Secondary Outcome: Remission Induction Rate After 2 Courses of Induction Therapy
Description: Patients without an evaluable bone marrow at the end of Induction I will be excluded from the calculation of remission rate after 2 courses of therapy because their responses are not evaluable. The following patients will be considered to not be in complete remission (CR) after 2 courses of therapy: (1) patients who die during Induction I and II; (2) patients with ≥ 5% blasts or extramedullary disease at the end of Induction II.
Time Frame: After 2 courses of induction (I and II) therapy, assessed for up to 10 years
Population: Ineligible (n=42) patients are excluded. Patients without an evaluable bone marrow at the end of Induction I or at the end of Induction II are excluded from the calculation of remission rate after 2 courses of therapy because their responses are not evaluable (n=45).
Measure: Number; unit: Proportion of participants
Arm/Group | Arm A: Standard Arm - No GMTZ, AML Pts w/Out Down Syndrome | Arm B: Experimental - With GMTZ, AML Pts w/Out Down Syndrome | Arm A: Standard Arm - No GMTZ, AML Patients With Down Syndrome
Number analyzed (Participants) | 491 | 486 | 6
Proportion of participants | 0.851324 | 0.882716 | 0.666667

4. Secondary Outcome: Disease-free Survival (DFS)
Description: Time from end of Intensification I to relapse, death or last contact
Time Frame: At 3 years from end of Intensification I
Population: Ineligible (n=42) patients are excluded. Patients who did not continue on therapy at end of Intensification I are also excluded (n=247).
Measure: Number (95% Confidence Interval); unit: Percentage participants DFS at 3 years
Arm/Group | Arm A: Standard Arm - No GMTZ, AML Pts w/Out Down Syndrome | Arm B: Experimental - With GMTZ, AML Pts w/Out Down Syndrome | Arm A: Standard Arm - No GMTZ, AML Patients With Down Syndrome
Number analyzed (Participants) | 377 | 400 | 4
Percentage participants DFS at 3 years | 56.6 [51.3 to 61.5] | 63.0 [58.0 to 67.5] | 75.0 [12.8 to 96.1]

5. Secondary Outcome: Mortality
Description: Number of participants who died during the first three courses of therapy.
Time Frame: During the first three courses of therapy
Population: Ineligible (n=42) patients are excluded.
Measure: Number; unit: Number of participants
Arm/Group | Arm A: Standard Arm - No GMTZ, AML Pts w/Out Down Syndrome | Arm B: Experimental - With GMTZ, AML Pts w/Out Down Syndrome | Arm A: Standard Arm - No GMTZ, AML Patients With Down Syndrome
Number analyzed (Participants) | 511 | 511 | 6
Number of participants | 11 | 13 | 1

6. Secondary Outcome: Time to Marrow Recovery
Description: Mean time to ANC recovery - defined as ANC greater than 500/MicroLiter for 3 consecutive days.
Time Frame: At 25 days after treatment with Induction I, Induction II, and Intensification I
Population: Excluded: Ineligible patients (pts) (n=42) for overall number of pts analyzed. For Induction I: Pts who did not have ANC recovery (n=237) or w/unknown (w/unk) status (n=14). For Induction II: Pts who did not have ANC recovery (n=142) or w/unk status (n=82). For Intensification I: Pts who did not have ANC recovery (n=104) or w/unk status (n=182)
Measure: Mean (Standard Deviation); unit: Mean days
Arm/Group | Arm A: Standard Arm - No GMTZ, AML Pts w/Out Down Syndrome | Arm B: Experimental - With GMTZ, AML Pts w/Out Down Syndrome | Arm A: Standard Arm - No GMTZ, AML Patients With Down Syndrome
Number analyzed (Participants) | 511 | 511 | 6
Mean days
  During Induction I (days 0 - 28 of therapy): number analyzed (Participants) | 380 | 391 | 6
  During Induction I (days 0 - 28 of therapy) | 30.56 (6.96) | 30.56 (6.47) | 29.17 (2.79)
  During Induction II (days 29 - 56 of therapy): number analyzed (Participants) | 394 | 405 | 5
  During Induction II (days 29 - 56 of therapy) | 28.54 (6.69) | 28.52 (6.25) | 26.6 (4.83)
  During Intensification I (days 57 - 84 of therapy): number analyzed (Participants) | 355 | 383 | 4
  During Intensification I (days 57 - 84 of therapy) | 27.51 (5.95) | 28.10 (6.32) | 24.5 (3.70)

7. Secondary Outcome: Toxicities, Including Infectious Complications
Description: Number of participants with at least one grade 3 or higher adverse event during therapy.
Time Frame: From the time therapy is initiated, assessed up to 10 years
Population: Ineligible (n=42) patients are excluded.
Measure: Number; unit: Number of participants
Arm/Group | Arm A: Standard Arm - No GMTZ, AML Pts w/Out Down Syndrome | Arm B: Experimental - With GMTZ, AML Pts w/Out Down Syndrome | Arm A: Standard Arm - No GMTZ, AML Patients With Down Syndrome
Number analyzed (Participants) | 511 | 511 | 6
Number of participants | 482 | 477 | 5

ADVERSE EVENTS:
Description: SAE field contains NCI Common Terminology Criteria for Adverse Events (CTCAEs) submitted via expedited reporting (NCI AdEERs / CAeRs). The AE field contains grade 3 and higher CTCAEs reported on study excluding those that were reported as SAEs. Ineligible patients are excluded from reporting of adverse events.
Arm/Group | Arm A: Standard Arm - No GMTZ, AML Pts w/Out Down Syndrome | Arm B: Experimental - With GMTZ, AML Pts w/Out Down Syndrome | Arm A: Standard Arm - No GMTZ, AML Patients With Down Syndrome
Serious Adverse Events (participants affected / at risk) | 26/511 | 32/511 | 2/6
Other Adverse Events (participants affected / at risk) | 482/511 | 479/511 | 5/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Standard Arm - No GMTZ, AML Pts w/Out Down Syndrome (N=511) | Arm B: Experimental - With GMTZ, AML Pts w/Out Down Syndrome (N=511) | Arm A: Standard Arm - No GMTZ, AML Patients With Down Syndrome (N=6)
Acidosis (Metabolism and nutrition disorders) | 3 | 3 | 0
Acute kidney injury (Renal and urinary disorders) | 8 | 2 | 0
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 4 | 8 | 0
Alanine aminotransferase increased (Investigations) | 0 | 2 | 0
Ascites (Gastrointestinal disorders) | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 2 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Atrial flutter (Cardiac disorders) | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 2 | 1 | 0
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Cardiac disorders - Other (Cardiac disorders) | 3 | 4 | 0
Confusion (Psychiatric disorders) | 0 | 1 | 0
Creatinine increased (Investigations) | 0 | 1 | 0
Death NOS (General disorders) | 3 | 3 | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 2 | 2 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 1 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 2 | 0
Fibrinogen decreased (Investigations) | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0
Heart failure (Cardiac disorders) | 1 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 2 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 6 | 4 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 7 | 7 | 2
Infections and infestations - Other (Infections and infestations) | 14 | 15 | 1
Intracranial hemorrhage (Nervous system disorders) | 0 | 6 | 0
Investigations - Other (Investigations) | 1 | 1 | 0
Left ventricular systolic dysfunction (Cardiac disorders) | 2 | 5 | 0
Lipase increased (Investigations) | 0 | 1 | 0
Lung infection (Infections and infestations) | 0 | 0 | 1
Mucositis oral (Gastrointestinal disorders) | 1 | 0 | 0
Multi-organ failure (General disorders) | 6 | 2 | 0
Nervous system disorders - Other (Nervous system disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 1 | 0
Pericarditis (Cardiac disorders) | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Pleural hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0
Portal hypertension (Hepatobiliary disorders) | 1 | 0 | 0
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Restrictive cardiomyopathy (Cardiac disorders) | 1 | 0 | 0
Right ventricular dysfunction (Cardiac disorders) | 1 | 0 | 0
Seizure (Nervous system disorders) | 1 | 1 | 1
Sepsis (Infections and infestations) | 1 | 2 | 0
Serum amylase increased (Investigations) | 0 | 1 | 0
Sudden death NOS (General disorders) | 1 | 1 | 0
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Vascular disorders - Other (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Standard Arm - No GMTZ, AML Pts w/Out Down Syndrome (N=511) | Arm B: Experimental - With GMTZ, AML Pts w/Out Down Syndrome (N=511) | Arm A: Standard Arm - No GMTZ, AML Patients With Down Syndrome (N=6)
Abdominal distension (Gastrointestinal disorders) | 3 | 4 | 0
Abdominal infection (Infections and infestations) | 2 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 38 | 44 | 0
Abducens nerve disorder (Nervous system disorders) | 0 | 2 | 0
Acidosis (Metabolism and nutrition disorders) | 7 | 13 | 0
Activated partial thromboplastin time prolonged (Investigations) | 13 | 15 | 0
Acute kidney injury (Renal and urinary disorders) | 9 | 25 | 1
Adrenal insufficiency (Endocrine disorders) | 0 | 2 | 0
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 21 | 37 | 0
Agitation (Psychiatric disorders) | 2 | 4 | 0
Alanine aminotransferase increased (Investigations) | 84 | 103 | 0
Alkaline phosphatase increased (Investigations) | 0 | 2 | 0
Alkalosis (Metabolism and nutrition disorders) | 2 | 4 | 0
Allergic reaction (Immune system disorders) | 0 | 0 | 1
Anal mucositis (Gastrointestinal disorders) | 5 | 3 | 0
Anal pain (Gastrointestinal disorders) | 7 | 7 | 0
Anal ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Anaphylaxis (Immune system disorders) | 25 | 32 | 1
Anemia (Blood and lymphatic system disorders) | 10 | 8 | 0
Anorectal infection (Infections and infestations) | 0 | 4 | 0
Anorexia (Metabolism and nutrition disorders) | 144 | 165 | 2
Anxiety (Psychiatric disorders) | 2 | 3 | 0
Apnea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0
Arachnoiditis (Nervous system disorders) | 1 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 2 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 18 | 19 | 0
Aspartate aminotransferase increased (Investigations) | 55 | 73 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0
Ataxia (Nervous system disorders) | 3 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Avascular necrosis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 14 | 11 | 0
Bladder infection (Infections and infestations) | 6 | 4 | 0
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 1 | 1 | 0
Blood bilirubin increased (Investigations) | 57 | 61 | 0
Blurred vision (Eye disorders) | 2 | 2 | 0
Bone infection (Infections and infestations) | 1 | 2 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 3 | 0
Bronchial infection (Infections and infestations) | 1 | 2 | 0
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 | 5 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 0
Burn (Injury, poisoning and procedural complications) | 0 | 1 | 0
Buttock pain (Musculoskeletal and connective tissue disorders) | 2 | 4 | 0
Capillary leak syndrome (Vascular disorders) | 0 | 3 | 0
Cardiac arrest (Cardiac disorders) | 2 | 2 | 0
Cardiac disorders - Other (Cardiac disorders) | 110 | 95 | 1
Cardiac troponin T increased (Investigations) | 0 | 1 | 0
Catheter related infection (Infections and infestations) | 2 | 4 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 1 | 0
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0
Chills (General disorders) | 2 | 3 | 0
Cholecystitis (Hepatobiliary disorders) | 4 | 2 | 0
Chronic kidney disease (Renal and urinary disorders) | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 18 | 9 | 0
Colonic fistula (Gastrointestinal disorders) | 1 | 0 | 0
Colonic hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Confusion (Psychiatric disorders) | 4 | 4 | 0
Conjunctivitis (Eye disorders) | 1 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 6 | 0
CPK increased (Investigations) | 1 | 1 | 0
Creatinine increased (Investigations) | 13 | 9 | 0
Cystitis noninfective (Renal and urinary disorders) | 1 | 5 | 0
Cytokine release syndrome (Immune system disorders) | 2 | 3 | 0
Death NOS (General disorders) | 1 | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 16 | 16 | 0
Dental caries (Gastrointestinal disorders) | 0 | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 3 | 4 | 0
Depression (Psychiatric disorders) | 6 | 3 | 0
Diarrhea (Gastrointestinal disorders) | 80 | 58 | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 8 | 13 | 0
Dizziness (Nervous system disorders) | 1 | 2 | 0
Duodenal hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 2 | 0
Dysphagia (Gastrointestinal disorders) | 4 | 3 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 22 | 24 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 0
Edema face (General disorders) | 0 | 1 | 0
Edema limbs (General disorders) | 1 | 1 | 0
Edema trunk (General disorders) | 3 | 1 | 0
Electrocardiogram QT corrected interval prolonged (Investigations) | 69 | 68 | 0
Encephalopathy (Nervous system disorders) | 5 | 5 | 0
Endocrine disorders - Other (Endocrine disorders) | 1 | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 2 | 2 | 0
Enterocolitis infectious (Infections and infestations) | 20 | 19 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 16 | 23 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Esophageal hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Esophageal pain (Gastrointestinal disorders) | 3 | 2 | 0
Esophagitis (Gastrointestinal disorders) | 12 | 12 | 0
Euphoria (Psychiatric disorders) | 1 | 0 | 0
External ear pain (Ear and labyrinth disorders) | 0 | 1 | 0
Eye disorders - Other (Eye disorders) | 2 | 1 | 0
Eye infection (Infections and infestations) | 0 | 3 | 0
Eye pain (Eye disorders) | 1 | 5 | 0
Facial nerve disorder (Nervous system disorders) | 0 | 2 | 0
Facial pain (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 7 | 4 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 267 | 280 | 4
Fever (General disorders) | 26 | 21 | 0
Fibrinogen decreased (Investigations) | 7 | 3 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Gallbladder infection (Infections and infestations) | 1 | 0 | 0
Gallbladder necrosis (Hepatobiliary disorders) | 1 | 0 | 0
Gallbladder obstruction (Hepatobiliary disorders) | 2 | 1 | 0
Gallbladder pain (Hepatobiliary disorders) | 1 | 0 | 0
Gastric hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 9 | 3 | 0
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 3 | 8 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 1 | 0
General disorders and administration site conditions - Other (General disorders) | 9 | 2 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0
GGT increased (Investigations) | 25 | 41 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 2 | 0
Glucose intolerance (Metabolism and nutrition disorders) | 1 | 1 | 0
Gum infection (Infections and infestations) | 0 | 3 | 0
Headache (Nervous system disorders) | 19 | 28 | 0
Hearing impaired (Ear and labyrinth disorders) | 1 | 0 | 0
Heart failure (Cardiac disorders) | 2 | 1 | 0
Hematoma (Vascular disorders) | 1 | 2 | 0
Hematuria (Renal and urinary disorders) | 3 | 6 | 0
Hemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0 | 0
Hepatic pain (Hepatobiliary disorders) | 13 | 16 | 0
Hepatobiliary disorders - Other (Hepatobiliary disorders) | 1 | 1 | 0
Hydrocephalus (Nervous system disorders) | 1 | 0 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 2 | 3 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 117 | 124 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 25 | 39 | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 5 | 14 | 0
Hypernatremia (Metabolism and nutrition disorders) | 7 | 16 | 1
Hypertension (Vascular disorders) | 22 | 38 | 0
Hypertriglyceridemia (Metabolism and nutrition disorders) | 3 | 6 | 0
Hyperuricemia (Metabolism and nutrition disorders) | 2 | 7 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 24 | 24 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 56 | 44 | 1
Hypoglycemia (Metabolism and nutrition disorders) | 3 | 4 | 0
Hypokalemia (Metabolism and nutrition disorders) | 169 | 191 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 17 | 9 | 0
Hyponatremia (Metabolism and nutrition disorders) | 59 | 63 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 43 | 58 | 0
Hypotension (Vascular disorders) | 80 | 79 | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 77 | 84 | 1
Ileus (Gastrointestinal disorders) | 7 | 9 | 0
Immune system disorders - Other (Immune system disorders) | 1 | 0 | 0
Infections and infestations - Other (Infections and infestations) | 395 | 406 | 4
Infective myositis (Infections and infestations) | 1 | 0 | 0
Injury, poisoning and procedural complications - Other (Injury, poisoning and procedural complications) | 0 | 1 | 0
INR increased (Investigations) | 5 | 5 | 0
Insomnia (Psychiatric disorders) | 3 | 0 | 0
Intra-abdominal hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Intracranial hemorrhage (Nervous system disorders) | 2 | 2 | 0
Intraoperative gastrointestinal injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Intraoperative respiratory injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Investigations - Other (Investigations) | 5 | 0 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Kidney infection (Infections and infestations) | 1 | 0 | 0
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
Left ventricular systolic dysfunction (Cardiac disorders) | 32 | 21 | 0
Lip infection (Infections and infestations) | 0 | 1 | 0
Lip pain (Gastrointestinal disorders) | 2 | 0 | 0
Lipase increased (Investigations) | 27 | 21 | 0
Localized edema (General disorders) | 1 | 0 | 0
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 4 | 5 | 0
Lung infection (Infections and infestations) | 12 | 9 | 0
Lymph gland infection (Infections and infestations) | 0 | 3 | 0
Malabsorption (Gastrointestinal disorders) | 0 | 1 | 0
Meningitis (Infections and infestations) | 0 | 1 | 0
Middle ear inflammation (Ear and labyrinth disorders) | 1 | 2 | 0
Mucosal infection (Infections and infestations) | 1 | 1 | 0
Mucositis oral (Gastrointestinal disorders) | 82 | 94 | 2
Multi-organ failure (General disorders) | 0 | 3 | 0
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 6 | 0
Myocarditis (Cardiac disorders) | 1 | 1 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Nausea (Gastrointestinal disorders) | 49 | 62 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Nervous system disorders - Other (Nervous system disorders) | 0 | 2 | 0
Neuralgia (Nervous system disorders) | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 15 | 11 | 0
Non-cardiac chest pain (General disorders) | 7 | 6 | 0
Oculomotor nerve disorder (Nervous system disorders) | 0 | 1 | 0
Oral hemorrhage (Gastrointestinal disorders) | 3 | 1 | 0
Oral pain (Gastrointestinal disorders) | 28 | 35 | 0
Otitis media (Infections and infestations) | 0 | 1 | 0
Pain (General disorders) | 15 | 20 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 12 | 15 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 2 | 4 | 0
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 2 | 0
Pancreatitis (Gastrointestinal disorders) | 4 | 3 | 0
Paroxysmal atrial tachycardia (Cardiac disorders) | 2 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 1 | 0 | 0
Penile infection (Infections and infestations) | 0 | 2 | 0
Penile pain (Reproductive system and breast disorders) | 0 | 2 | 0
Pericardial effusion (Cardiac disorders) | 8 | 4 | 1
Pericarditis (Cardiac disorders) | 0 | 1 | 0
Perineal pain (Reproductive system and breast disorders) | 2 | 3 | 0
Peripheral motor neuropathy (Nervous system disorders) | 2 | 4 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 3 | 6 | 0
Personality change (Psychiatric disorders) | 1 | 0 | 0
Pharyngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 5 | 5 | 0
Pharyngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 0 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 | 8 | 0
Photophobia (Eye disorders) | 3 | 4 | 0
Platelet count decreased (Investigations) | 13 | 12 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 19 | 16 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 39 | 29 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Portal hypertension (Hepatobiliary disorders) | 7 | 6 | 0
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 2 | 1 | 0
Proctitis (Gastrointestinal disorders) | 1 | 0 | 0
Proteinuria (Renal and urinary disorders) | 2 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 4 | 0
Psychosis (Psychiatric disorders) | 6 | 3 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 0
Purpura (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 25 | 29 | 0
Rectal fistula (Gastrointestinal disorders) | 1 | 0 | 0
Rectal hemorrhage (Gastrointestinal disorders) | 2 | 0 | 0
Rectal mucositis (Gastrointestinal disorders) | 2 | 1 | 0
Rectal pain (Gastrointestinal disorders) | 14 | 9 | 0
Renal and urinary disorders - Other (Renal and urinary disorders) | 3 | 3 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 7 | 5 | 0
Restrictive cardiomyopathy (Cardiac disorders) | 4 | 1 | 0
Rhinitis infective (Infections and infestations) | 1 | 0 | 0
Right ventricular dysfunction (Cardiac disorders) | 2 | 0 | 0
Scrotal infection (Infections and infestations) | 0 | 2 | 0
Seizure (Nervous system disorders) | 7 | 5 | 0
Sepsis (Infections and infestations) | 4 | 8 | 0
Serum amylase increased (Investigations) | 16 | 8 | 0
Sinus bradycardia (Cardiac disorders) | 2 | 1 | 0
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Sinus tachycardia (Cardiac disorders) | 6 | 10 | 0
Sinusitis (Infections and infestations) | 1 | 3 | 0
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 3 | 5 | 0
Skin induration (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Skin infection (Infections and infestations) | 10 | 7 | 0
Skin ulceration (Skin and subcutaneous tissue disorders) | 3 | 3 | 0
Small intestinal mucositis (Gastrointestinal disorders) | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 1 | 0
Small intestine infection (Infections and infestations) | 3 | 2 | 0
Soft tissue infection (Infections and infestations) | 2 | 7 | 0
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Stomach pain (Gastrointestinal disorders) | 3 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 2 | 1 | 0
Syncope (Nervous system disorders) | 5 | 9 | 0
Thromboembolic event (Vascular disorders) | 3 | 9 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 3 | 1 | 0
Tracheal hemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0
Tracheitis (Infections and infestations) | 1 | 0 | 0
Tumor lysis syndrome (Metabolism and nutrition disorders) | 9 | 9 | 0
Typhlitis (Gastrointestinal disorders) | 29 | 31 | 0
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 3 | 0
Upper respiratory infection (Infections and infestations) | 5 | 8 | 0
Urinary frequency (Renal and urinary disorders) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 11 | 8 | 0
Urinary tract obstruction (Renal and urinary disorders) | 2 | 0 | 0
Urinary tract pain (Renal and urinary disorders) | 2 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 3 | 2 | 0
Uterine hemorrhage (Reproductive system and breast disorders) | 2 | 6 | 0
Uterine pain (Reproductive system and breast disorders) | 0 | 1 | 0
Uveitis (Eye disorders) | 0 | 1 | 0
Vaginal hemorrhage (Reproductive system and breast disorders) | 1 | 6 | 0
Vaginal infection (Infections and infestations) | 1 | 0 | 0
Vaginal pain (Reproductive system and breast disorders) | 1 | 1 | 0
Vascular access complication (Injury, poisoning and procedural complications) | 5 | 5 | 0
Vascular disorders - Other (Vascular disorders) | 5 | 5 | 0
Vasculitis (Vascular disorders) | 1 | 1 | 0
Venous injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 2 | 4 | 0
Vitreous hemorrhage (Eye disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 34 | 44 | 0
Vulval infection (Infections and infestations) | 1 | 0 | 0
Weight gain (Investigations) | 16 | 16 | 0
Weight loss (Investigations) | 21 | 12 | 0
White blood cell decreased (Investigations) | 11 | 8 | 0
Wound infection (Infections and infestations) | 4 | 4 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Must obtain prior Sponsor approval.